CLINICAL TRIAL: NCT00409149
Title: Comprehensive Approach to Lower Measured Blood Pressure (CALM-BP) - Results From a Randomized Controlled Trial
Brief Title: The Effect of a Complementary Multi Disciplinary Program on Blood Pressure in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 140/06
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2007-04

CONDITIONS: Hypertension
Keywords: Hypertension; Diet; physical exercise; naturopathic; group therapy; Qi Gong
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CALM BP (Experimental): dietary approach, education on cooking and food consumption choices, walking physical exercise, Qi Gong - a form of Chinese slow movement exercise combined with relaxation breathing and imagery and group therapy coaching in stress management techniques and mind-body balancing techniques.
  Interventions: Behavioral: CALM Approache
- DASH (Active Comparator): standard dietary DASH approach in hypertensive patients
  Interventions: Behavioral: DASH approach

INTERVENTIONS:
Behavioral: CALM Approache
  Arms: CALM BP
Behavioral: DASH approach — standard dietary DASH approach in hypertensive patients
  Arms: DASH

SUMMARY:
Intervention description:

Complementary Approaches to Lower Mean arterial pressure (CALM) is a multi dispensary program aimed to reduce blood pressure in hypertensive patients. The program utilizes a naturopathic dietary approach, education on cooking and food consumption choices, walking physical exercise, Qi Gong - a form of Chinese slow movement exercise combined with relaxation breathing and imagery and group therapy coaching in stress management techniques and mind-body balancing techniques.

Trial Objectives:

To compare the effect of CALM in reducing blood pressure to the standard dietary DASH approach in hypertensive patients.

Methodology:

120 Participants will be randomly assigned in to two groups:

* CALM program for reducing blood pressure as the treatment group.
* Standard DASH diet and lifestyle modification counseling as the control group. Inclusion Criteria
* Adult men and women over 18 years.
* Patients using anti hypertensive medications with mean systolic blood pressure measurements of 120-180 mm Hg and/or mean diastolic measurements of 70-100 mm Hg as determined by a 24 hour Holter test.
* Patients not using anti hypertensive medications with mean systolic blood pressure measurements of 130-180 mm Hg and or mean diastolic measurements of 80-100 mmHg.
* Signed informed consent (appears in IRB forms)

Assessment of Efficacy Primary end point efficacy will be assessed by comparing the mean BP measurements in the CALM group to the mean BP measurements in the DASH control group. Blood pressure measurements will be performed by 24 hours Holter BP monitoring in the beginning and at the end of the trial.

Secondary end points efficacy will be assed by comparing CALM to DASH programs with respect to effects use of BP medications and weight loss. Lab test and pulse wave analysis will also be assessed at the beginning and at the end of the study.

DETAILED DESCRIPTION:
Intervention description Complementary Approaches to Lower Mean arterial pressure (CALM) utilizes a naturopathic dietary approach, education on cooking and food consumption choices, walking physical exercise, Qi Gong - a form of Chinese slow movement exercise combined with relaxation breathing and imagery and group therapy coaching in stress management techniques and mind-body balancing techniques.

Trial Objectives

Primary objective To compare the effect of CALM in reducing blood pressure to the standard dietary DASH approach in hypertensive patients.

Secondary objectives To provide information on the efficacy of CALM in reducing weight and improving quality of life. and to examine it's potential to indicate a dose reduction in hypertensive medications. To evaluate CALM effects on cardiovascular disease risk factors.

Trial Design

A single center parallel randomized control trial including two groups and enrolling 120 participants.

Primary End Point A comparable change in blood pressure measurements between CALM and DASH groups after the 16 week period of the trial as measured by a 24 hour holter test which will be performed in the beginning and the end of the study.

Secondary End Points

A comparable change in hypertensive medications A comparable change in weight reduction

Comparable changes in cardiovascular risk factors as indicated by following laboratory tests and evaluations :

Arterial wall thickening , hemoglobin, hemoglobin A1c, creatinine, liver function parameters, highly sensitive c-reactive protein (hsCRP), low density lipoprotein (LDL), high density lipoprotein (HDL), triglycerides (TG), oxidized LDL (oxLDL), nitric oxide metabolites and microalbumine/creatinine ratio.

Methodology 120 Participants will be randomly assigned in to two groups:

* CALM program for reducing blood pressure as the treatment group.(As described below in section 6)
* Standard DASH diet and lifestyle modification counseling as the control group. (As described below in section 6)

Duration of the study Group intervention in the treatment arm consists of 16 weeks of the CALM program. Due to the limited number of participants we can allocate to each group, three 16 weeks cycles will be repeated in order to recruit the needed number of participants for the trial. Thus the treatment phase is expected to last for 48 weeks. Recruitment is expected to last about three months. An additional 6 months will be required for completion of data entry and analysis.

Location of the study The study will take place in Asaf Harofeh Medical Center, Israel and will be conducted in Shiram - The Department of Integrated Medicine and in the Research and Development Unit of Assaf Harofeh Medical Center.

Recruitment of the Subjects Patients will be recruited from the community and from Asaf Harofeh medical center. Patients from a number of departments within the hospital will be invited to participate in the study. An advertisement in the local newspaper and in the medical center's web site will be published (appears in IRB forms) Recruitment will continue until the overall quota of subjects (50 per group) will be met.

Randomization Subjects will be randomly assigned to each treatment group utilizing a computerized randomization system. A random list will be generated by the study statistician. The random list will be kept in a sealed envelope in the study site. The list will be readily available in case of any emergency.

Follow up Subjects will be assessed in the beginning and at the end of the trial and again 6 months later. Compliance questioners will be filled during several stages of the trial as described in section 8 below.

Study Population Inclusion Criteria

* Adult men and women over 18 years.
* Patients using anti hypertensive medications with mean systolic blood pressure measurements of 120-180 mm Hg and/or mean diastolic measurements of 70-100 mm Hg as determined by a 24 hour Holter test.
* Patients not using anti hypertensive medications with mean systolic blood pressure measurements of 130-180 mm Hg and or mean diastolic measurements of 80-100 mmHg.
* Signed informed consent Exclusion Criteria
* Cardiovascular event within the past 6 months
* Inability to walk independently for 15 or less minutes.
* Poorly controlled insulin dependant diabetes mellitus with Hg A1c measurements over 7.5.
* Inflammatory bowl disorders
* Acute malignancy with life expectancy of less than 5 years.
* Pregnancy or lactation
* A body mass index of more than 35.
* More than 20 alcoholic beverages per weak.
* Change in anti hypertensive medications within the last 3 months.
* Planning to change smoking habits

Treatment of the subjects

The CALM group will receive a weekly 4 hour group coaching session for 16 weeks. Each session will include the following parts:

1. A group aerobic walking session. Participants will reach a target heart rate which will be determined in advance as 60-75% of maximal heart rate expected for their age and with accordance to their physical ability. The group walk will last for a maximum of one hour. All participants will be encouraged to walk at least 3 times per week independently.

   .
2. A 1 hour weekly Qi Gong session. The class will include 45 minutes of slow movement exercises emphasizing relaxation, abdominal breathing and visualization stretching and meditation. A 15 minutes prerecorded guided imagery meditation aimed to reduce blood pressure will be performed in a seated or supine position. Participants will be given a CD with the 15 minutes mediation and will be encouraged to use it at home once a day.
3. Dietary counseling and cooking instructions for forming a healthy home cooking routine which will be based on naturopathic rice diet approach. A group meal will be prepared by participants in each session and participants will dine together. All participants will be encouraged to follow the same diet at home.
4. Group therapy meeting focusing on stress management techniques and mind - body balancing. Emphasis will be put on developing communication skills based on nonjudgmental and empathic approaches, methods for dealing with stress and anxiety, discarding low self esteem and negative thought patterns and developing positive thinking patterns.

The DASH control group will receive group coaching sessions for 16 weeks. Each session will include the following parts:

1. A group aerobic walking session. Participants will reach a target heart rate which will be calculated in advance as 60-75% of maximal heart rate expected for their age. The group walk will last for a maximum of one hour. All participants will be encouraged to walk at least 3 times per week independently.
2. Dietary counseling and cooking instructions according to a standard DASH diet. This will include a diet rich in fruits, vegetables and low fat dairy products. A group meal will be prepared by participants in each session and participants will dine together. All the participant will be encouraged to follow the same diet at home.

Assessment of Efficacy

Primary end point efficacy will be assessed by comparing the mean BP measurements in the CALM group to the mean BP measurements in the DASH control group. Blood pressure measurements will be performed by 24 hours Holter BP monitoring in the beginning and at the end of the trial.

Secondary end points efficacy will be assed by comparing CALM to DASH programs with respect to effects use of BP medications and weight loss. Lab test and pulse wave analysis will also be assessed at the beginning and at the end of the study.

Pulse wave analysis Assessment of arterial stiffness will be performed, at baseline, at the end of 16 weeks of the trial and following 6 months, by a noninvasive technique using the commercially available SphygmoCor System (AtCor Medical,LTD, Australia). All measurements will be performed by S.E while the patient is in the recombinant position at room temperature of 25oc. In brief, peripheral pressure waveforms will be recorded from the radial artery at the wrist, using applanation tonometry with a high-fidelity micromanometer (Millar Instruments). When 20 sequential waveforms will be recorded, a validated 16-18 generalized transfer function will be applied to generate the corresponding central aortic pressure waveform. Augmentation index (AIx) and augmented pressure (AP) were derived by calculation, using pulse wave analysis technique. The merging point of the incident and the reflected wave (the inflection point) will be identified on the generated aortic pressure waveform. AP will be calculated as maximum systolic pressure minus pressure at the inflection point. AIx will be calculated as AP divided by pulse pressure and expressed as percentage. Higher values of AIx indicated increased wave reflection from the periphery or earlier return of the reflected wave as a result of increased pulse wave velocity (attributable to increased arterial stiffness), and vice versa. Only high-quality recordings, defined as those with in-device quality index >80% (as derived from an algorithm including average pulse height, pulse height variations, diastolic variations, and the maximum rate of rise of the peripheral waveform) and the curves acceptable upon a visual inspection performed by one investigator, will be included in the analysis. All pulse wave measurements will be taken in the same sitting position, in a quiet, temperature controlled room (23 ± 1°C), after at least 15 minute resting period.

Laboratory Tests At the beginning and at the end of the study, blood will be drawn for measurement of hemoglobin, hemoglobin A1c, creatinine, liver function tests, highly sensitive c-reactive protein (hsCRP) and lipid profile including total cholesterol high density lipoprotein (HDL) and triglycerides (TG). LDL will calculated. Five cc of plasma will be preserved in -70oc for future evaluation of oxidative stress (oxLDL, MDA) and NO.

Life Quality & well being questioners Patients will fill the MOS 36 life quality questionnaire in the beginning, at week 4, week 10 and at the end of the trial. In addition a specific questionnaire for assessing dietary and cooking lifestyle will be filled in the begging and at the end of the trial. These questionnaires will again be after six months for the follow up period.

Compliance Compliance questionnaires will address three topics: adherence to the diet recommendations and cooking instructions at home, number of exercise sessions per week and frequency of using the Qi Gong meditation disk at home. Questionnaires will be filled at the end of weeks 4,10 & 16 (end of trial) and at the follow up meeting post 6 months.

Assessment of Safety No adverse events or risks are expected for participants enrolled in this trial. However, initially, the strict dietary program may influence the participants overall energy level. Transient symptoms such as dizziness and headaches may also present in early stages of the study participants will be couched in advance on how to maintain any undesired influences. Nevertheless, any adverse event will be reported on the Adverse Event Form along with the probability of the adverse event being study-related.

Decreasing doses or cessation of BP Medications use BP medication doses will be changed by the primary investigator or by the patient healthcare physician. The physician in charge will reduce BP lowering medications in case systolic blood pressure will decrease below 110 mmHg or if participants will present symptoms of low blood pressure such as weakness, ortostatizm, dizziness, presyncope or syncope. Before any change in BP lowering medications patients will be encouraged to get another 24 hours holter of BP measurement test. All changes in BP medications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 18 years.
* Patients using anti hypertensive medications with mean systolic blood pressure measurements of 120-180 mm Hg and/or mean diastolic measurements of 70-100 mm Hg as determined by a 24 hour Holter test.
* Patients not using anti hypertensive medications with mean systolic blood pressure measurements of 130-180 mm Hg and or mean diastolic measurements of 80-100 mmHg.
* Signed informed consent

Exclusion Criteria:

* Cardiovascular event within the past 6 months
* Inability to walk independently for 15 or less minutes.
* Poorly controlled insulin dependant diabetes mellitus with Hg A1c measurements over 7.5.
* Inflammatory bowl disorders
* Acute malignancy with life expectancy of less than 5 years.
* Pregnancy or lactation
* A body mass index of more than 35.
* More than 20 alcoholic beverages per weak.
* Change in anti hypertensive medications within the last 3 months.
* Planning to change smoking habits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Principal Investigator — Assaf-Harofeh Medical Center; Amos Ziv, M.Sc., Study Chair — Assaf-Harofeh Medical Center
Locations (1):
- Research & Development Unit, Assaf-Harofeh Medical Center,, Ẕerifin, Israel